CLINICAL TRIAL: NCT05711238
Title: The Effect of Robotic Hand Therapy on Hand Functions and Quality of Life in Children With Cerebral Palsy: A Randomized Controlled Study
Brief Title: Robotic Hand Therapy for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, assistant professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SASPHAND
Record Dates: First submitted 2023-01-09; First posted 2023-02-02 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy; Hand Functions; Rehabilitation; Robotic Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot Assisted Therapy Group (Experimental): Investigators planned to apply robotic rehabilitation therapy with a hand-finger robot [Amadeo (Tyromotion, Graz, Austria)] for 40 minutes, accompanied by a physiotherapist who is trained in the field of robotic rehabilitation and has at least 5 years of experience for the hands on the affected side of the children in the Robot Assisted Therapy Group group.
  Amadeo (Tyromotion, Graz, Austria) is an end-effector device designed for the hand. It is a groove-shaped device attached to the forearm using magnets using bandages on the fingers.
  Interventions: Other: Robotic rehabilitation; Other: Conventional rehabilitation
- Conventional Therapy Group (Active Comparator): Conventional therapy group In the pediatric rehabilitation of the children's hands on the affected side, an exercise program consisting of 40 minutes of hand finger joint range of motion exercises (passive, active assistive), strengthening exercises, and coarse and fine dexterity exercises was planned, accompanied by a physiotherapist experienced for at least 5 years.
  A total of 30 sessions of treatment were planned for both groups, 5 days a week. It will be recommended that they continue with the same dose of the medical treatment they have been using during the treatment program. Children will be evaluated by a physiatrist blinded to groups before and after treatment.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Robotic rehabilitation — In robot-assisted therapy, the therapist selects different programs with personalized environments to train patients to strengthen limb muscles that have previously had difficulty with movements or are relatively weak. Active (individual finger movement, memory, motility, apple tree, target board, recycling bins, balloons, firefighter), auxiliary, and passive (cpm, cpm plus) treatment options are available in the system.
  Arms: Robot Assisted Therapy Group
Other: Conventional rehabilitation — Conventional therapy group In the pediatric rehabilitation of the children's hands on the affected side, an exercise program consisting of 40 minutes of hand finger joint range of motion exercises (passive, active assistive), strengthening exercises, and coarse and fine dexterity exercises was planned, accompanied by a physiotherapist experienced for at least 5 years.

SUMMARY:
Cerebral palsy (CP) is the most common physical disability in childhood. The term CP is defined as a group of persistent but non-progressive movement and posture disorders resulting from a defect or lesion of the immature brain. The overall prevalence of CP worldwide is 2.11 per 1000 live births.

There is evidence that 80% of children with CP have upper extremity involvement. In general, the acquisition of effective arm and hand skills for use in daily life is a complex process that not only requires neuromusculoskeletal integrity, but also includes various aspects of the child's abilities. Thus, in addition to the positive symptoms that typically present patterns of spasticity, children and adolescents with CP often have a poor ability to reach, grasp, release, and manipulate objects. They also have difficulty using their upper extremities to perform self-care and other activities.

Robot-assisted and computer-assisted methods may be valuable new strategies for improving the sensory-motor learning process in children with central motor impairment. These new technologies represent an attractive complement to existing physiotherapeutic and occupational therapy concepts.

In patients with difficulty in individual finger and hand movements, the AMADEO device (Tyromotion, Austria) can be used for unilateral distal training of the upper extremity. With this device, patients with little or no voluntary control of the hand and fingers can receive more or less passive training, while those with better distal function of the upper extremity can strength train by following the device or even against the device to a certain extent.

Implementation of robot-assisted therapy provides intense repetitive training, sensorimotor integration and cognitive engagement through targeted tasks; focuses primarily on functional motor performance. From previous studies, the use of robotic devices has been found to improve the kinematics, range of motion, muscle tone, postural control, and functionality of the upper and lower extremities in individuals with CP. Robotic hand therapy has started to take place in routine rehabilitation protocols today. Considering the scarcity of studies on robotic hand therapy in the pediatric group, larger-scale studies are needed. In this study, our aim is to investigate the effect of robotic hand therapy on hand functions and quality of life in children with CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common physical disability in childhood. The term CP is defined as a group of persistent but non-progressive movement and posture disorders resulting from a defect or lesion of the immature brain. The overall prevalence of CP worldwide is 2.11 per 1000 live births.

There is evidence that 80% of children with CP have upper extremity involvement. In general, the acquisition of effective arm and hand skills for use in daily life is a complex process that not only requires neuromusculoskeletal integrity, but also includes various aspects of the child's abilities. Thus, in addition to the positive symptoms that typically present patterns of spasticity, children and adolescents with CP often have a poor ability to reach, grasp, release, and manipulate objects. They also have difficulty using their upper extremities to perform self-care and other activities.

Robot-assisted and computer-assisted methods may be valuable new strategies for improving the sensory-motor learning process in children with central motor impairment. These new technologies represent an attractive complement to existing physiotherapeutic and occupational therapy concepts.

In patients with difficulty in individual finger and hand movements, the AMADEO device (Tyromotion, Austria) can be used for unilateral distal training of the upper extremity. With this device, patients with little or no voluntary control of the hand and fingers can receive more or less passive training, while those with better distal function of the upper extremity can strength train by following the device or even against the device to a certain extent.

Implementation of robot-assisted therapy provides intense repetitive training, sensorimotor integration and cognitive engagement through targeted tasks; focuses primarily on functional motor performance. From previous studies, the use of robotic devices has been found to improve the kinematics, range of motion, muscle tone, postural control, and functionality of the upper and lower extremities in individuals with CP.

In a case series of 7 children with CP presenting the results of robotic therapy, it showed beneficial effects on body structure and function, including motor function, coordination, and brachioradial muscle recruitment, but no improvement in activity and participation skills. It has been stated that there is a need for new studies to be carried out with longer training periods and with the measurement of grip strength, daily living activity evaluation scales covering a wide variety of tasks.

In the first randomized controlled study with 16 children with CP, the results of upper extremity robot-assisted therapy were evaluated with body functions, structure and activity participation scales, and it was found that robotic therapy improved upper extremity kinematics and manual dexterity, but not functional activities and social participation.

Most robotic studies in children and adolescents with CP have relatively small sample sizes and few randomized controlled trials.

Robotic hand therapy has started to take place in routine rehabilitation protocols today. Considering the scarcity of studies on robotic hand therapy in the pediatric group, larger-scale studies are needed. In this study, our aim is to investigate the effect of robotic hand therapy on hand functions and quality of life in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* grade 1-3 according to the manual ability classification system
* capable of taking multi-step commands
* able to sit in a chair

Exclusion Criteria:

* Having persistent pain in the upper extremity or hand (VAS>40)
* with severe spasticity of the hand (MAS≥3) or contracture
* Fracture or operation in the upper extremity in the past 6 months
* Botulinum toxin injection to the upper extremity in the last 6 months
* skin ulcer
* severe vision and hearing impairment
* intense ataxia
* uncontrolled epilepsy

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
MACS (Manual Ability Classification System for Children with Cerebral Palsy) | 15 minutes
  It is designed to classify how children with CP aged 4-18 use their hands while manipulating objects in daily life. The starting point of MACS is in upper extremity function, but it is also influenced by environmental, personal and contextual factors. It is designed to reflect the child's typical manual performance. MACS is a five-level system where level I represents the best dexterity and level V indicates that the child is not using their hands for functional purposes. It is intended to indicate the level that best represents the child's usual performance at home, school, and community settings. The Turkish version of the MACS has been found to be valid and reliable and is recommended to be suitable for the assessment of manual dexterity in the Turkish population.
Spasticity Evaluation | 5 minutes
  It was planned to evaluate spasticity with the Modified Ashworth Scale (MAS). In MAS, patients are evaluated over 5 points. 0; there is no increase in muscle tone, and 4 indicates that the extremity is rigid in flexion and extension.

SECONDARY OUTCOMES:
Jamar Dynamometer | 5 minutes
  Measurements will be made with the shoulder adjacent to the trunk in adduction and neutral rotation, elbow 90 degrees flexed, wrist 0-30 degrees dorsiflexion and 0-15 degrees ulnar deviation with thumbs up. In the hand on the affected side, the measurements will be repeated three times with an interval of 5 seconds, and the average of the three measurements will be recorded in kilograms. Finger grip strength will be evaluated with a 'Jamar digital pinchmeter'. Patients will be placed in a sitting position with the wrist in 90° flexion and the forearm in a neutral position. Measurements will be made bilaterally in three different positions as lateral, palmar and fingertip grips. Patients will be asked to squeeze with maximum force and each measurement will be made three times, and their averages will be recorded in kg.
Jebsen Taylor Hand Function Test | 45 minutes
  The test is used in the age range of 6 - 90 years. Test items
  1 - Card flip (measuring 3x 5 inches) 2- Collecting small objects and throwing them into cans (2 paper clips, 2 coins and 2 soda caps) 3 - Stacking the backgammon pieces on top of each other (wooden backgammon pieces are used) 4- Writing (24-word sentence) Jumping 5-5 light cans across 6- Jumping 5 heavy tin cans across 7 - Collecting 5 dried kidney beans using a teaspoon Among the test materials, the commands to be used during the test are written in detail in the user manual of the test. Test supplies include a scale board to ensure a standard arrangement of objects used, and a stopwatch to measure the time the activities are performed. If the child fails the activity, that part of the test is not continued.
Box Block Test | 75 minutes
  Box Block Test Dexterity is evaluated with the box-block test. KBT consists of a wooden box divided into two compartments by 150 blocks. In CBT, the person being tested is asked to move the blocks in one compartment to the other compartment as quickly as possible within 60 seconds. The test is started with the dominant hand and the test is repeated with both hands. There is also a 15 second trial period for both hands. The test is started by holding the blocks in the compartment on the side of the hand to be tested and positioning the box so that it is on the midline of the person being tested. When the time expires, the moved blocks are counted and the result is recorded (74). Validity and reliability studies of CBT were conducted.
Nine Hole Peg Test | 30 minutes
  Nine Hole Peg Test This test measures dexterity based on performance (in seconds). A wooden board with nine holes on it, 9 short wooden sticks and a box in which the wooden sticks can be placed are placed in front of the patient. Using the hand to be evaluated, the patient is asked to place the wooden sticks in the box into the holes on the panel as quickly as possible, and then put the sticks back into the box one by one. The completion time of the test is determined by the stopwatch.
ABILHAND- Kids Manual Ability Scale | 30 minutes
  ABILHAND Kids survey of the child; It is used to assess dexterity, defined as the ability to manage daily activities that require the use of the upper extremities, regardless of the strategies involved. The questionnaire, consisting of 18 items, including unimanual and bimanual activities, is answered by the parents of the children with a 3-level scale (0 cannot do one activity, 1 activity is difficult, 2 activities are easily done).
Pediatric Functional Independence Measurement | 30 minutes
  Pediatric Functional Independence Measurement (WeeFIM) measures children's level of functional independence in activities of daily living. Evaluation is done with the participation of parents. In total, 18 activities consisting of 6 main headings are questioned, and a score between 1 and 7 is given for each activity. The highest score that can be obtained is 126, while the lowest score is 18 points. Validity and reliability studies of the (WeeFIM) for Turkey have been carried out.
Quality of Life Scale for Children - SP Module (PedsQL-CP) | 30 minutes
  The 35-item PedsQL 3.0 SP Module consists of seven subscales: Daily Activities (9 items), School Activities (4 items), Movement and Balance (5 items), Pain and Pain (4 items), Fatigue (4 items), Eating Activities (5 topics), Speech and Communication (4 topics). The scale consists of a child self-report report and a parent report. Child self-report reports include ages 5-7 (young), ages 8-12 (child), and ages 13-18 (young). Parental reports include ages 2-4 (infant), ages 5-7 (young), ages 8-12 (child), and ages 13-18 (young), and assess parents' perceptions of their child's health-related quality of life. The scale questions the degree of problems children have experienced in the last month.
Fugl Meyer Upper Extremity Assessment Questionnaire | 15 minutes
  The Fugl-Meyer Upper Extremity Motor Rating Scale was developed to quantitatively evaluate sensorimotor recovery after stroke. Based on Brunnstrom's stages of motor recovery. FMUE Scale consists of 33 items, each scored from 0 to 2. where 0 = unable to perform, 1 = partially performs and 2 = fully performs. The total score is 66. Higher scores indicate better motor functions.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA ADAR, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Sevda Adar, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Derived] Adar S, Keskin D, Dundar U, Toktas H, Yesil H, Eroglu S, Eyvaz N, Bestas E, Demircan A. Effect of Robotic Rehabilitation on Hand Functions and Quality of Life in Children With Cerebral Palsy: A Prospective Randomized Controlled Study. Am J Phys Med Rehabil. 2024 Aug 1;103(8):716-723. doi: 10.1097/PHM.0000000000002430. Epub 2024 Jan 31. PMID 38320248